CLINICAL TRIAL: NCT06063746
Title: Compassionate Use of Vidutolimod
Status: No longer available | Type: Expanded Access
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CMP-001-Vidutolimod
Record Dates: First submitted 2023-09-18; First posted 2023-10-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Refractory Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Vidutolimod
  Other Names: CMP-001

SUMMARY:
Provide Compassionate Use of Vidutolimob

DETAILED DESCRIPTION:
Compassionate use is only available to patients who transitioned from a previous vidutolimod (CMP-001) study.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult